CLINICAL TRIAL: NCT07128836
Title: Effects of Insole Vibration With Proprioceptive Training on Balance and Functional Ability in Patients With Diabetic Peripheral Nuropathy
Brief Title: Effects of Insole Vibration With Proprioceptive Training in Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0263 Rabia Shahzadi
Record Dates: First submitted 2025-04-17; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Peripheral Neuropathy (DPN)
Keywords: Diabetic polyneuropathy; Vibrating insole,; Proprioceptive training; Balance
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Vibration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants in this arm will perform both proprioceptive training exercises and receive insole vibrator.
  Interventions: Other: proprioceptive training exercise and receive insole vibrator
- Group B (Active Comparator): Participants in this arm will receive only proprioceptive training exercise along with simple insoles without vibration.
  Interventions: Other: proprioceptive training exercise along with simple insoles without vibration

INTERVENTIONS:
Other: proprioceptive training exercise and receive insole vibrator — The treatment for the participants in the experimental group includes; 5 minutes warm up, 30 minutes proprioceptive training exercise, 20 minutes walk with in-sole vibrator, 5 minutes cool down. The duration of each session will be 60 minutes. All the participants will receive 36 sessions (3 times per week over 12 week's period).
  Arms: Group A
Other: proprioceptive training exercise along with simple insoles without vibration — The treatment for the participants in the control group includes; 5 minutes warm up, 30 minutes proprioceptive training exercise, 20 minutes walk with non-vibrating insole, 5 minutes cool down. The duration of each session will be 60 minutes. All the participants will receive 36 sessions (3 times per week over 12 week's period).
  Arms: Group B

SUMMARY:
Diabetic peripheral neuropathy (DPN) is a prevalent complication of diabetes, profoundly affecting quality of life with sensory disturbances and associated complications. Proprioceptive training shows promise in improving proprioception and functional outcomes in patients with peripheral neuropathy. Also the literature has shown that Insole vibrator demonstrates potential in mitigating symptoms and improving sensory function and balance in patients with peripheral neuropathy. This study aims to determine the effects of insole vibration with proprioceptive training on balance and functional ability in patient with diabetic peripheral neuropathy.

In this randomized controlled trial design, 60 participants will be recruited. The sample size was calculated through G-power total of 60 participants. Who meet the inclusion criteria will be recruited through non-probability convenience sampling technique, which will further be randomized through online randomizer tool into control and experimental group with thirty participants in each group. Experimental group will receive proprioceptive training alongside vibrating insole and control group will receive proprioceptive training with non vibrating insoles. Data will be collected by using various assessment tools, including Numeric Pain Rating Scale for pain,Time Up And Go Test for functional mobility, Neuropathic Disability Score for level of disability ,Functional Reach Test for standing stability, Mini BESTS for balance, functional mobility and gait, Single Leg Stance Test for static posture and balance control and the Montreal Cognitive Assessment for cognitive impairment. Pre-intervention assessments will be conducted for both groups. The effects of the interventions will be measured at pre-treatment, 6th week, 12th week and at 16th week. Data analysis will be performed by using SPSS 26. Mixed ANOVA and repeated-measures ANOVA will use for within-group analysis whereas between-group analysis will perform by using one-way ANOVA.

Key words: Diabetic polyneuropathy, Vibrating insole, proprioceptive training, balance

ELIGIBILITY:
Inclusion Criteria:

* • Patients with both genders male and female will be included

  * The age limit for the patients will be from 50 to 70 years
  * Patients diagnosed with DPN type 1 or type 2
  * Patients with neuropathic disability score greater than 3 will be included
  * Patients with Michigan questionnaire higher than 3
  * Patients who can walk independently with BBS score between 41 to 56

Exclusion Criteria:

* Patients with Mini Mental State less than 24
* Patients having Numeric Pain Rating Scale greater than 4
* Patients with any impairment in lower leg e.g; Leg Length Discrepancy, foot ulcer, lower limb injury

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline after completion of 6 and 8 weeks
  to measure pain scale range 0-10. zero means no pain 10 means maximum
Time Up and Go (TUG) Test | Baseline after completion of 6 and 8 weeks
  To measure mobility and fall risk (time to rise, walk, return) measure in seconds time > 20 sec means impaired mobility
Neuropathic Disability score (NDS) | Baseline after completion of 6 and 8 weeks
  Severity of PND (0-10 scale) 0 means no disability 10 means maximum disability
Functional Reach test (FRT) | Baseline after completion of 6 and 8 weeks
  to measure anticipatory postural control Stability and fall risk
Mini-BESTest | Baseline after completion of 6 and 8 weeks
  to measure static and dynamic balance (0-30 scale) greater score means better mobility

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- Chiniot General Hospital and Civil Hospital (Allied 2), Faisalabad, Faisalābad, Pakistan

IPD SHARING:
Plan to Share IPD: No